CLINICAL TRIAL: NCT05167786
Title: Locomotor Function Following Transcutaneous Electrical Spinal Cord Stimulation in Individuals With Hemiplegic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00215009
Record Dates: First submitted 2021-12-07; First posted 2021-12-22 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Aim 1: Gait Training + Stimulation (Experimental): Up to 60 min of locomotion training with transcutaneous spinal cord stimulation. However, the amount of time spent in side-lying locomotion training, treadmill training and over ground training will depend on individual tolerance and progression.
  Interventions: Device: Noninvasive spinal stimulation with gait training; Other: Exploratory Phase - Optimization of Gait Training and Spinal Stimulation
- Aim 1: Gait Training + Sham Stimulation (Active Comparator): Up to 30 seconds of transcutaneous spinal cord stimulation in order to blind them to the intervention while performing locomotion training. However, the amount of time spent in side-lying locomotion training, treadmill training and over ground training will depend on individual tolerance and progression.
  Interventions: Device: Conventional gait training
- Aim 2: Gait Training + Stimulation (Experimental): Up to 60 min of locomotion training with transcutaneous spinal cord stimulation. However, the amount of time spent in side-lying locomotion training, treadmill training and over ground training will depend on individual tolerance and progression.
  Interventions: Device: Noninvasive spinal stimulation with gait training; Other: Exploratory Phase - Optimization of Gait Training and Spinal Stimulation
- Aim 2: Gait Training + Sham Stimulation (Active Comparator): Up to 30 seconds of transcutaneous spinal cord stimulation in order to blind them to the intervention while performing locomotion training. However, the amount of time spent in side-lying locomotion training, treadmill training and over ground training will depend on individual tolerance and progression.
  Interventions: Device: Conventional gait training

INTERVENTIONS:
Device: Noninvasive spinal stimulation with gait training — Transcutaneous Spinal Cord Neurostimulator will deliver transcutaneous electrical spinal cord stimulation while subjects perform lower limb locomotor activities.
  Arms: Aim 1: Gait Training + Stimulation; Aim 2: Gait Training + Stimulation
Device: Conventional gait training — Subjects will receive lower limb locomotion training without transcutaneous spinal cord stimulation. However, the amount of time spent in side-lying locomotion training, treadmill training and over ground training will depend on individual tolerance and progression.
  Arms: Aim 1: Gait Training + Sham Stimulation; Aim 2: Gait Training + Sham Stimulation
Other: Exploratory Phase - Optimization of Gait Training and Spinal Stimulation — Subjects may receive various lower limb locomotion training with or without transcutaneous spinal cord stimulation. Training approaches may include but are not limited to single or split belt treadmill and over ground walking. Transcutaneous Spinal Cord Neurostimulator may deliver a variety of transcutaneous electrical spinal cord stimulation to subjects.
  Arms: Aim 1: Gait Training + Stimulation; Aim 2: Gait Training + Stimulation

SUMMARY:
This study has two interventional components, the first is a cross-over design and the second is a randomized control trial. Both will evaluate the effectiveness of transcutaneous (non-invasive) spinal cord stimulation on gait and balance function for individuals with hemiplegia due to stroke.

DETAILED DESCRIPTION:
OBJECTIVES:

* Exploratory phase: Identify a systematic, methodical approach to identifying the optimal stimulation parameters and gait training protocol for each individual patient with stroke.
* Aim 1: Evaluate short-term effects of transcutaneous spinal cord stimulation + gait training on gait symmetry, gait performance, and corticospinal circuitry in individuals with chronic stroke.
* Aim 2: Evaluate and predict long-term effects of transcutaneous spinal cord stimulation + gait training on gait symmetry, gait performance, and corticospinal circuitry in individuals with chronic stroke
* Aim 3: Identify parameters that distinguish responders from non-responders to transcutaneous spinal cord stimulation in individuals with chronic stroke.

ELIGIBILITY:
Inclusion Criteria

* Age 18 years or older
* Able and willing to give written consent and comply with study procedures
* At least 6 months' post-stroke
* Hemiplegia secondary to a single stroke
* Functional Ambulation Category of 2 or greater - i.e., subject needs continuous or intermittent support of one person to help with balance and coordination.
* Not currently receiving regular physical therapy services
* Physician approval to participate

Exclusion Criteria

* Ataxia
* Multiple stroke history
* Botox injection in lower extremity within the last 4 months
* Modified Ashworth score of 3 or greater in lower extremity
* Pregnant or nursing
* Using a powered, implanted cardiac device for monitoring or support of heart function (i.e. pacemaker, defibrillator, or LVAD) or anti-spasticity implantable pumps
* Active pressure sores
* Unhealed bone fractures
* Peripheral neuropathies
* Painful musculoskeletal dysfunction due to active injuries or infections
* Severe contractures in the lower extremities
* Medical illness limiting the ability to walk
* Active urinary tract infection
* Clinically significant depression, psychiatric disorders, or ongoing drug abuse
* Active cancer or cancer in remission less than 5 years
* Orthopedic dysfunction, injury, or surgery that would impact an individual's ability to use the lower extremity.
* Traumatic brain injury or other neurological conditions that would impact the study.

TMS-Specific Exclusion Criteria: TMS will be utilized for both Aims. The sub-set of participants who meet these criteria will participate in this component of the studies.

* Medicated with agents known to increase (e.g., amphetamines) or decrease motor system excitability (e.g., lorazepam)
* Implanted cardiac pacemaker
* Metal implants in the head or face
* Suffers unexplained, recurring headaches
* Had a seizure in the past unrelated to the stroke event, or has epilepsy
* Skull abnormalities or fractures
* A concussion within the last 6 months
* Unstable cardiorespiratory or metabolic diseases (e.g. cardiac arrhythmia, uncontrolled hypertension, uncontrolled diabetes, or chronic emphysema)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-08-25 (Estimated); Study Completion 2027-08-25 (Estimated)

PRIMARY OUTCOMES:
Change in Gait Symmetry | Aim 1: Baseline pre-intervention immediately post intervention for interventions 1, 2, 3 and 4. Aim 2: Baseline pre-intervention, 4 weeks into the intervention, immediately post intervention and 3 months post intervention for intervention 1 and 2.
  Participants will ambulate along Gait Rite electronic walkway 3 times per gait speed to evaluate gait pattern at both their self-selected and safe fast gait speed. The GAITRite electronic walkway contains sensor pads encapsulated in a carpet and connected to a computer. The system can be laid over any flat surface and automates measuring temporal and spatial gait parameters. The GAITRite electronic walkway for the study shall be a minimum of 14 feet long. The GAITRite data capture was chosen as measurement of the patient's overall gait quality.

SECONDARY OUTCOMES:
Change in 6 Minute Walk Test | Aim 2: Baseline pre-intervention, 4 weeks into the intervention, immediately post intervention and 3 months post intervention for intervention 1 and 2.
  The 6 Minute Walk Test (6MWT) measures the distance a subject can walk indoors on a flat, hard surface in a period of 6 minutes, using assistive devices, as necessary. The test is a reliable and valid evaluation of functional exercise capacity and is used as a sub-maximal test of aerobic capacity and endurance. The test will be used to determine participant's gait efficiency at baseline and at study completion. The walk test is patient self-paced and assesses the level of functional capacity. Patients are allowed to stop and rest during the test, however, the timer does not stop. If the patient is unable to complete the time, the time stopped is noted and reason for stopping prematurely is recorded.
  This test will be administered while wearing a portable gas analysis system called the Cosmed K4B2 to measure oxygen consumption. This system measures oxygen consumption (VO2) and Carbon-dioxide production (VCO2) in a breath by breath fashion.
Change in 10 Meter Walk Test | Aim 1: Baseline pre-intervention immediately post intervention for interventions 1, 2, 3 and 4. Aim 2: Baseline pre-intervention, 4 weeks into the intervention, immediately post intervention and 3 months post intervention for intervention 1 and 2.
  This test will examine the patient's gait speed. Patients will be directed to walk 3 times per gait speed to evaluate gait pattern at both their self-selected and safe fast gait speed. Patients will be positioned 1 meter before the start line and instructed to walk the entire distance and past the end line approximately 1 meter. The distance before and after the course are meant to minimize the effect of acceleration and deceleration. Time will be recorded using a stopwatch and recorded to the one hundredth of a second (ex: 2.15 sec).

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States